CLINICAL TRIAL: NCT05641493
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of HLX208 （BRAF V600E Inhibitor） Combined With Serplulimab（HLX10, Anti-PD-1 Antibody） in Advanced NSCLC Patients With BRAF V600E Mutation.
Brief Title: A Phase Ib/II Clinical Trial to Evaluate the Safety and Efficacy of HLX208+HLX10 in NSCLC With BRAF V600E Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-NSCLC203
Record Dates: First submitted 2022-11-15; First posted 2022-12-07 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: HLX208; HLX10; BRAF V600E mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX208 combined HLX10 (Experimental): For the phase Ib study, HLX208 is administered orally at two dose levels of 600mg BID or 900 mg BID. And HLX10 is administered intravenously at a fixed dose of 300mg every 3 weeks.
  For the phase II study, HLX208 is administered orally with the RP2D dose. And HLX10 is administered intravenously at a fixed dose of 300mg every 3 weeks.
  Interventions: Combination Product: HLX208+HLX10

INTERVENTIONS:
Combination Product: HLX208+HLX10 — HLX208 is a BRAF V600E inhibitor ,and HLX10 is an anti-PD-1 monoclonal antibody.

SUMMARY:
An open-label, multicenter phase Ib/II clinical study to evaluate safety, tolerability, pharmacokinetics, and efficacy of HLX208 (BRAF V600E Inhibitor) combined with HLX10 （anti-PD-1 monoclonal antibody）in advanced NSCLC patients with BRAF V600 mutation.

DETAILED DESCRIPTION:
This is an open-label, multicenter phase Ib/II clinical study to evaluate safety, tolerability, pharmacokinetics, and efficacy of HLX208 (BRAF V600E Inhibitor) combined with HLX10 （anti-PD-1 monoclonal antibody）in advanced NSCLC patients with BRAF V600 mutation.

For the phase Ib study, HLX208 is administered orally at two dose levels of 600mg BID or 900 mg BID. And HLX10 is administered intravenously at a fixed dose of 300mg every 3 weeks.

For the phase II study, HLX208 is administered orally with the RP2D dose. And HLX10 is administered intravenously at a fixed dose of 300mg every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤75 years old of age (in phase Ib study) or ≥18 and ≤80 years old of ag (in phase II study) at the time of informed consent.
2. Signed written informed consent.
3. BRAF V600E mutant advanced solid tumors (in phase Ib study) or advanced NSCLC (in phase II study) patients with positive PD-L1 expression (TPS or TC≥1%).
4. Previous failure of standard therapy, intolerance to standard therapy, lack of standard therapy, or currently unsuitable for standard therapy.
5. Prior systemic anti-neoplastic therapy (chemotherapy, radiotherapy, targeted therapy, or traditional Chinese medicine with anti-neoplastic indications) must have been ≥ 2 weeks from the first dose in this study with treatment-related AE resolved to NCI-CTCAE Grade ≤ 1 (except for alopecia)
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
7. Expected survival time ≥ 3 months.
8. At least one measurable target lesion per RECIST v1.1 (brain metastasis could not be considered as the only measurable lesion).
9. With normal major organ functions (no blood transfusions or treatment with colony-stimulating factor within 14 days prior to the first dose in this study).
10. Be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bow
11. Fertile subjects (male or female) must agree to take effective contraceptive measures from the time of signing the ICF until 90 days after the last dose of HLX208 or 6 months after the last dose of HLX10. Female subjects of childbearing potential must complete a pregnancy test with a negative result within 7 days prior to the first dose.

Exclusion Criteria:

1. For subjects in phase II study: previous treatment with BRAF inhibitors or MEK inhibitors or previous treatment with T cell co-stimulation or immune checkpoint therapy.
2. Known EGFR mutations or ALK rearrangements (except in subjects with EGFR mutations whose disease has progressed after previous EGFR inhibitor treatment).
3. Received strong CYP3A inhibitors or inducers treatment within 1 week prior to the first dose of investigational product.
4. Received major surgery within 28 days prior to the first dose of investigational product. A major surgery is defined as a surgery that takes at least 3 weeks of postoperative recovery before receiving treatment in this study.
5. With uncontrolled pleural effusion, pericardial effusion, or ascites.
6. With symptomatic brain or meningeal metastases (unless the patient has been treated for >3 months, there is no evidence of progression on imaging within 4 weeks prior to the first dose, and the tumor-related clinical symptoms are stable).
7. With active pulmonary tuberculosis. Patients with previous and current interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, or severe impaired pulmonary function that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
8. With any serious infection requiring systemic anti-infective therapy within 14 days prior to the first dose of the investigational product.
9. History of other malignant tumors (except for cured carcinoma in situ of the cervical or basal cell carcinoma of the skin) within two years prior to the first dose of investigational product.
10. Being positive (+) for hepatitis B surface antigen (HBsAg) or positive (+) for hepatitis B core antibody (HBcAb), and with hepatitis B virus deoxyribonucleic acid (HBV-DNA) ≥ 2500 copies/mL or 500 IU/mL.
11. Being positive (+) for HCV RNA.
12. Being positive (+) human immunodeficiency virus (HIV) antibody.
13. History of serious cardiovascular and cerebrovascular diseases.
14. Systemic treatment with corticosteroids (> 10 mg/day prednisone or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of the investigational product or during the study. In the absence of active autoimmune disease, subjects are allowed to use inhaled or topical steroids, or adrenal hormone replacement therapy at an effective dose equivalent to ≤10 mg/day prednisone.
15. Known active or suspected autoimmune diseases. Subjects with autoimmune related hypothyroidism receiving thyroid hormone replacement therapy are allowed to participate in the study. Subjects with stable type 1 diabetes receiving insulin therapy are allowed to participate in the study.
16. Known alcohol of or drug abuse.
17. Pregnant or lactating women.
18. Received live vaccine within 28 days prior to the first dose of investigational product.
19. Have other conditions not suitable for inclusion as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-03-04 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
MTD (for phase Ib study) | From first dose to the end of Cycle 1 (each cycle is 3 weeks).
  The maximum tolerated dose of HLX208 combined with HLX10.
DLT (for phase Ib study) | From first dose to the end of Cycle 1 (each cycle is 3 weeks).
  The proportion of patients experiencing dose limiting toxicity (DLT) events.
ORR (for phase II study) | up to approximately up to 24 months
  Objective response rate assessed by the investigator per RECIST 1.1.

SECONDARY OUTCOMES:
PFS | approximately up to 36 months
  Progression-Free-Survival
DCR | approximately up to 24 months
  Disease-Control-Rate
DOR | approximately up to 24 months
  Duration of Overall Response
TTR | approximately up to 24 months
  Time to Tumor Response
12-month OS rate | 12 months
  12-month OS rate
6-month OS rate | 6 months
  6-month OS rate
OS | approximately up to 48 months
  Overall-Survival
12-month PFS rate | 12 months
  12-month PFS rate
6-month PFS rate | 6 months
  6-month PFS rate
SAE | approximately up to 48 months
  The proportion of patients experiencing SAE.
AUC0-T | From First administration of HLX 208 to 12 weeks.
  Area under the concentration-time curve from time 0 to the last concentration measurable time point.
AUC0-∞ | From First administration of HLX 208 to 12 weeks.
  Area under the concentration-time curve from time 0 to infinity.
Cmax | From First administration of HLX 208 to 12 weeks.
  Peak Plasma Concentration.
Tmax | From First administration of HLX 208 to 12 weeks.
  Time to first occurrence of Cmax
t1/2 | From First administration of HLX 208 to 12 weeks.
  Elimination half-life
AUCss | From First administration of HLX 208 to 12 weeks.
  Area under the steady-state concentration-time curve

OTHER OUTCOMES:
Association of biomarkers with efficacy | approximately up to 48 months
  Association of efficacy with biomarkers including PD-L1 expression, BRAF V600E mutation abundance, MSI status and TMB status.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Dr., Principal Investigator — Shanghai Chest Hospital, Shanghai Jiao Tong University School Of Medicine
Locations (1):
- Shanghai Chest Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No